CLINICAL TRIAL: NCT06764485
Title: A Phase 3, Two-part, Randomized, Open-label, Adaptive Study Comparing BMS-986365 Versus Investigator's Choice of Therapy Comprising Either Docetaxel or Second Androgen Receptor Pathway Inhibitor (ARPI), in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) - rechARge
Brief Title: A Study to Compare the Efficacy and Safety of BMS-986365 Versus the Investigator's Choice of Therapy in Participants With Metastatic Castration-resistant Prostate Cancer
Acronym: rechARge
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA071-1000; 2024-517422-25 (Other: EU CTR); U1111-1311-0532 (Other: WHO)
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate cancer; Protein degrader; Protein degradation; Androgen receptor; Castrate resistant prostate cancer; Castration resistant prostate cancer; Hormone resistant; Metastatic hormone resistant prostate cancer; Metastatic castrate resistant prostate cancer; Metastatic castration resistant prostate cancer; BMS-986365; CC-94676; CA071-1000; CA0711000; rechARge; Abiraterone; Docetaxel; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — enzalutamide; abiraterone; Docetaxel; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: Dose 1 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Dose 2 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Comparator 1 (Active Comparator): Enzalutamide or Abiraterone Acetate + Prednisone/Prednisolone
  Interventions: Drug: Enzalutamide; Drug: Abiraterone; Drug: Predinsone/Prednisolone
- Part 1: Comparator 2 (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: Predinsone/Prednisolone
- Part 2: Dose Selected (Experimental)
  Interventions: Drug: BMS-986365
- Part 2: Comparator 1 (Active Comparator): Enzalutamide or Abiraterone Acetate + Prednisone/Prednisolone
  Interventions: Drug: Enzalutamide; Drug: Abiraterone; Drug: Predinsone/Prednisolone
- Part 2: Comparator 2 (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: Predinsone/Prednisolone

INTERVENTIONS:
Drug: BMS-986365 — Specified dose on specified days
  Arms: Part 1: Dose 1; Part 1: Dose 2; Part 2: Dose Selected
Drug: Enzalutamide — Specified dose on specified days
  Arms: Part 1: Comparator 1; Part 2: Comparator 1
Drug: Abiraterone — Specified dose on specified days
  Arms: Part 1: Comparator 1; Part 2: Comparator 1
Drug: Docetaxel — Specified dose on specified days
  Arms: Part 1: Comparator 2; Part 2: Comparator 2
Drug: Predinsone/Prednisolone — Specified dose on specified days
  Arms: Part 1: Comparator 1; Part 1: Comparator 2; Part 2: Comparator 1; Part 2: Comparator 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of BMS-986365 versus the investigator's choice of therapy in participants with Metastatic Castration-resistant Prostate Cancer.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to assess the radiographic progression free survival (rPFS) of BMS-986365 versus investigator's choice comprising Docetaxel + Prednisone/Prednisolone or Abiraterone + Prednisone/Prednisolone or Enzalutamide.

In Part 1, participants will be randomized 1:1:1 to one of the two BMS-986365 dose levels, or to the active comparator arm (investigator's choice). In Part 2 of the study, participants will be randomized 1:1 between BMS-986365 selected dose, or to the active comparator arm (investigator's choice).

ELIGIBILITY:
Inclusion Criteria

* Participants must have histologic or cytologic confirmation of adenocarcinoma of the prostate without small cell or neuro-endocrine features.
* Participants must have current evidence of metastatic disease documented by either bone lesions on radionuclide bone scan and/or soft tissue lesions on computed tomography/magnetic resonance imaging (CT/MRI).
* Participants must be asymptomatic or mildly symptomatic from prostate cancer with score on Brief Pain Inventory - Short Form (BPI-SF) that must be < 4.
* Participants must have had previous treatment with an androgen receptor pathway inhibitor (abiraterone, enzalutamide, apalutamide, or darolutamide).

Exclusion Criteria

* Participants must not have impaired cardiac function or clinically significant cardiac disease.
* Participants must not have any brain metastasis.
* Participants must not have any liver metastasis.
* Participants with superscan on technetium-99m (Tc-99m) radionuclide bone scans.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 960 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-09-12 (Estimated); Study Completion 2029-01-19 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) by blinded independent central review (BICR) using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (soft tissue) and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) (bone) criteria | Up to 4 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 4 years
Recommended dose of BMS-986365 for Part 2 | Up to approximately 1.5 years
Progression-free survival (PFS) | Up to 4 years
Confirmed overall response rate (ORR) by BICR assessment in participants with measurable disease using RECIST 1.1 (soft tissue) and PCWG3 (bone) criteria | Up to 4 years
Time to pain progression (TTPP) | Up to 4 years
Time to symptomatic progression (TTSP) | Up to 4 years
Time to initiation of the first subsequent systemic therapy (TFST) | Up to 4 years
Prostate-specific antigen (PSA) response rate | Up to 4 years
Change from baseline in Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P) total scores | Up to 4 years
Change from baseline in Prostate Cancer Subscale (PCS) scores | Up to 4 years
Change from baseline in trial outcome index (TOI) | Up to 4 years
Change from baseline in Brief Pain Inventory - Short Form (BPI-SF) worst pain (item #3) intensity | Up to 4 years
Incidence of adverse events (AEs) | Up to 4 years
Incidence of serious adverse events (SAEs) | Up to 4 years
Incidence of AEs leading to dose modifications | Up to 4 years
Incidence of AEs leading to interruptions | Up to 4 years
Incidence of AEs leading to discontinuation | Up to 4 years
Electrocardiogram (ECG) findings | Up to 4 years
  ECG Findings defined as :
  * Number of Postbaseline Abnormal Corrected QT (QTc) Values
  * Number of abnormal Beats Per Minute (BPM)
Incidence of laboratory abnormalities | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (279):
- United States (53):
  - Central Alabama Research, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Los Angeles Cancer Network (LACN), Anaheim, California
  - Moores Cancer Center, La Jolla, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Local Institution - 0364, Los Angeles, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - San Francisco VA Health Care System, San Francisco, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - Chesapeake Urology, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - James M Stockman Cancer Institute, Frederick, Maryland
  - Local Institution - 0104, Minneapolis, Minnesota
  - Local Institution - 0049, Las Vegas, Nevada
  - Thomas Jefferson University, Kennedy Health Alliance, Sewell, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants Ltd., Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Local Institution - 0085, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Associated Medical Professionals - Urology, Syracuse, New York
  - Local Institution - 0056, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Local Institution - 0433, Allentown, Pennsylvania
  - Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Urology Austin, PLLC, Austin, Texas
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Local Institution - 0220, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Local Institution - 0023, Richmond, Virginia
  - Local Institution - 0078, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (8):
  - Hospital Británico de Buenos Aires, CABA, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, ABB, Buenos Aires F.D.
  - Hospital Italiano de Córdoba, Córdoba, Córdoba Province
  - Local Institution - 0130, Río Cuarto, Córdoba Province
  - Clinica Viedma S. A, Viedma, R
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Hospital Privado Universitario de Córdoba, Córdoba
- Australia (16):
  - GenesisCare - Campbelltown, Campbelltown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - Port Macquarie - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Greenslopes Private Hospital - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital - Malvern, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (4):
  - Universitätsklinikum Krems, Krems, Lower Austria
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Brazil (6):
  - Local Institution - 0039, Vitória, Espírito Santo
  - Cetus Oncologia - Unidade Belo Horizonte, Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sírio Libanês, São Paulo, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
- Canada (9):
  - BC Cancer Kelowna, Kelowna, British Columbia
  - BC Cancer Vancouver, Vancouver, British Columbia
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Sunnybrook Research Institute, Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski, Rimouski, Quebec
- Chile (4):
  - Oncocentro Valdivia, Valdivia, Los Ríos Region
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Fundacion Arturo Lopez Perez (FALP), Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (39):
  - Second Affiliated hospital of Anhui Medical University, Hefei, Anhui
  - Local Institution - 0168, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Local Institution - 0176, Beijing, Beijing Municipality
  - Local Institution - 0237, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Local Institution - 0415, Huizhou, Guangdong
  - Local Institution - 0222, Harbin, Heilongjiang
  - Local Institution - 0211, Zhengzhou, Henan
  - Local Institution - 0279, Zhengzhou, Henan
  - Local Institution - 0284, Wuhan, Hubei
  - Local Institution - 0216, Changsha, Hunan
  - Local Institution - 0217, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Local Institution - 0228, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus), Nanchang, Jiangxi
  - Local Institution - 0198, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Local Institution - 0300, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Local Institution - 0212, Shanghai, Shanghai Municipality
  - Local Institution - 0215, Shanghai, Shanghai Municipality
  - Local Institution - 0308, Shanghai, Shanghai Municipality
  - Local Institution - 0205, Taiyuan, Shanxi
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - Local Institution - 0181, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Local Institution - 0280, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Local Institution - 0223, Wenzhou, Zhejiang
- Czechia (8):
  - Local Institution - 0011, Hořovice, Beroun
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Urocentrum Praha, Prague, Praha 2
  - Local Institution - 0418, Prague, Praha 4
  - Fakultni nemocnice v Motole, Prague, Praha 5
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (4):
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
- France (11):
  - Centre Antoine-Lacassagne, Nice, Alpes-Maritimes
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg, Alsace
  - Local Institution - 0432, Dijon, Côte-d'Or
  - Oncopole Claudius Regaud, Toulouse, Haute-Garonne
  - Local Institution - 0431, Saint-Grégoire, Ille-et-Vilaine
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy, Lorraine
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Clinique Victor Hugo Le Mans, Le Mans, Sarthe
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand
  - Local Institution - 0178, Paris
- Germany (14):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - TUM Klinikum, München, Bavaria
  - Local Institution - 0455, Bergisch Gladbach, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Local Institution - 0454, Biedenkopf
  - Universitätsklinikum Bonn, Bonn
  - Local Institution - 0456, Duisburg
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Marienhospital Herne, Herne
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- India (5):
  - Local Institution - 0404, Thiruvananthapuram, Kerala
  - Local Institution - 0401, Navi Mumbai, Maharashtra
  - Local Institution - 0402, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0400, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0405, Kolkata, West Bengal
- Ireland (3):
  - Cork University Hospital, Cork
  - Tallaght University Hospital, Dublin
  - Beaumont Hospital, Dublin, Dublin
- Italy (11):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Azienda USL 8 di Arezzo, Arezzo
  - Local Institution - 0424, Catania
  - Azienda Ospedaliero Universitaria Policlinico Riuniti di Foggia, Foggia
  - Local Institution - 0425, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - APSS- Presidio Ospedaliero S. Chiara, Trento
- Japan (19):
  - Local Institution - 0451, Nagoya, Aichi-ken
  - Local Institution - 0436, Sakura, Chiba
  - Local Institution - 0441, Matsuyama, Ehime
  - Local Institution - 0435, Sapporo, Hokkaido
  - Local Institution - 0446, Sapporo, Hokkaido
  - Local Institution - 0443, Kita-Gun, Kagawa-ken
  - Local Institution - 0444, Kamakura, Kanagawa
  - Local Institution - 0448, Yokohama, Kanagawa
  - Local Institution - 0437, Suita, Osaka
  - Local Institution - 0445, Bunkyo-ku, Tokyo
  - Local Institution - 0440, Koto-ku, Tokyo
  - Local Institution - 0438, Shinjuku-ku, Tokyo
  - Local Institution - 0447, Toyama, Toyama
  - Local Institution - 0450, Ube, Yamaguchi
  - Local Institution - 0439, Fukuoka
  - Local Institution - 0434, Kashiwa
  - Local Institution - 0449, Kobe
  - Local Institution - 0452, Kumamoto
  - Local Institution - 0442, Osaka
- Poland (8):
  - Pratia Poznań, Poznan, Greater Poland Voivodeship
  - POLIMED, Wroclaw, Lower Silesian Voivodeship
  - Państwowy Instytut Medyczny MSWiA, Warsaw, Masovian Voivodeship
  - SP ZOZ Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego w Opolu, Opole, Opole Voivodeship
  - COPERNICUS PL, Wojewodzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Regional Specialised Hospital No. 4 in Bytom, Bytom, Silesian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
- BRCR Global - Mayagüez, Mayagüez, Puerto Rico
- Romania (5):
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Spitalul Universitar C.F. Cluj-Napoca, Cluj-Napoca
  - Institutul Regional de Oncologie, Iași
  - Spitalul Municipal Schuller Ploiești, Ploieşti
- Slovakia (4):
  - MILAB, Prešov, Presov
  - Local Institution - 0275, Banská Bystrica
  - Local Institution - 0201, Bratislava
  - Local Institution - 0200, Martin, Žilina Region
- South Korea (6):
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (22):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona [Barcelona]
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo, Bizkaia
  - Local Institution - 0314, Santander, Cantabria
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital Lucus Augusti, Lugo, Lugo [Lugo]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense [Orense]
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de Burgos, Burgos
  - Hospital Vithas La Salud, Granada
  - Hospital Clinico San Carlos, Madrid
  - Local Institution - 0327, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (4):
  - Skånes Universitetssjukhus Lund, Lund, Skåne Län [se-12]
  - Karolinska Universitetssjukhuset Solna, Solna, Stockholms Län [se-01]
  - Akademiska sjukhuset, Uppsala, Uppsala Län [se-03]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands Län [se-14]
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (6):
  - Local Institution - 0340, Adana
  - Local Institution - 0339, Ankara
  - Local Institution - 0338, Ankara
  - Local Institution - 0341, Ankara
  - Local Institution - 0337, Istanbul
  - Local Institution - 0342, Istanbul
- United Kingdom (5):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Glasgow City
  - Mount Vernon Hospital, Northwood, Hillingdon
  - St Bartholomew's Hospital, London, London, City of
  - Royal Marsden Hospital (Sutton), London, Sutton
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Chi KN, McKay RR, Sandhu S, Arranz JA, Barthelemy P, Hadaschik B, Matsubara N, Shore ND, Ye D, Cascella T, Irincheeva I, Kreiser S, Thiery-Vuillemin A, Rathkopf DE. rechARge: a randomized phase III trial of the androgen receptor ligand-directed degrader, BMS-986365, vs investigator's choice in patients with mCRPC. Future Oncol. 2025 Jun;21(14):1771-1777. doi: 10.1080/14796694.2025.2502318. Epub 2025 Jun 2. PMID 40455815
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06764485.html